CLINICAL TRIAL: NCT00007358
Title: Study of Dexamethasone in Neonatal Lupus Congenital Heart Block; PRIDE (PR Interval and Dexamethasone Evaluation) in Congenital Heart Block
Brief Title: Dexamethasone Treatment for Congenital Heart Block (CHB) in Newborns With Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Jill Buyon, New York University Medical Center
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01AR046265 (NIH); R01AR046265 (NIH); NIAMS-055
Record Dates: First submitted 2000-12-19; First posted 2000-12-18 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Congenital Heart Block; Neonatal Lupus; Atrioventricular Nodal Dysfunction; Myocardial Injury
Keywords: Dexamethasone; Anti-SSA/Ro antibodies; Anti-SSB/La antibodies; Ultrasound; Atrioventricular (AV) nodal dysfunction; Echocardiograms; Mothers
MeSH Terms: conditions — Congenital heart block; Neonatal Systemic lupus erythematosus | interventions — Dexamethasone

ARMS (1):
- 1 (Experimental): Depending on patient and physician decision, a steroid may be administered during pregnancy.
  Interventions: Drug: Dexamethasone or other corticosteroid

INTERVENTIONS:
Drug: Dexamethasone or other corticosteroid — Administered during the third trimester of pregnancy

SUMMARY:
Some newborns are born with congenital heart block (CHB), a condition occurring in babies with neonatal lupus. The first part of the study will test the effectiveness of fluorinated steroids, including dexamethasone, in improving the heart function and general health of newborns who have auto-antibody-associated CHB. The second part of this study will use ultrasound and heart monitoring to observe high-risk pregnant women and their fetuses during the third trimester of pregnancy.

DETAILED DESCRIPTION:
CHB is an abnormal condition in which the heart beats slowly. This is a disease that is strongly associated with maternal antibodies to SSA/Ro and SSB/La ribonucleoproteins. This study hopes to clarify the causes of CHB and develop appropriate treatments. The study has two parts.

The first part of the study will be prospective; it will determine if fluorinated steroids given to women prior to birth improves the heart function and well-being of their newborns. This part of the study will evaluate fetuses diagnosed in utero with CHB during the third trimester of pregnancy. Diagnosis of CHB must occur at least 6 weeks before the baby is born to allow for sufficient data collection. It will be the decision of the physician and the mother as to whether a steroid will be administered. Fetuses will be evaluated before delivery by electrocardiogram (ECG) to detect abnormal fluid collection and by ultrasound to monitor heartbeat. After birth, newborns will be assessed for overall pumping strength of the heart and for abnormal heartbeat. Blood will be drawn from the mother at the time of enrollment and during delivery. Visits will occur over a span of approximately 5 months.

The second part of this study will be observational; the purpose is to identify classic indicators of heartbeat dysfunction and heart injury in newborns with CHB. The goal of this part of the study is to better understand the stages of heart injury, the role of anti-Ro/La antibodies in CHB, and procedures that may reverse heart block. Mothers considered to be at high risk for having a child with CHB will undergo weekly ECGs from 16 weeks into their pregnancy until Week 24, then will have an ECG every other week from Week 24 through Week 34. There will be a total of 15 visits to conduct these ECGs. Blood will be drawn at the first ECG visit and during delivery. Visits will occur over a span of 4 months.

For both parts of the study, babies will undergo ECGs after delivery and at one year of age. Additional tests not related to the study may be ordered by the physician.

ELIGIBILITY:
Inclusion Criteria for Prospective Part of Trial:

* Mother must have anti-Ro and/or anti-La antibody
* Fetal bradyarrhythmia (slow, abnormal heart rhythm)

Exclusion Criteria for Prospective Part of Trial:

* Fetal heart abnormalities that may cause newborn CHB and could account for atrioventricular (AV) block

Inclusion Criteria for Observational Part of Trial:

* Mother must have anti-Ro and/or anti-La antibody
* Fetus must have documented normal heartbeat prior to the 16th week of pregnancy
* Fetus must have a structurally normal heart
* Mother must be enrolled during the 16th, 17th, or 18th week of pregnancy

Exclusion Criteria for Observational Part of Trial:

* Mother is taking more than 10 mg of prednisone per day

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2000-10; Primary Completion 2007-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Neonatal ventricular heart rate | Measured over 5 months
Fractional shortening | Measured over 5 months
Abnormal fluid collection | Measured over 5 months

SECONDARY OUTCOMES:
Change in degree of heart block | Measured over 5 months
Gestational age (weeks) at birth | Measured over 5 months
Birth weight | Measured over 5 months
Cardiothoracic ratio | Measured over 5 months
EKG and echocardiogram | Measured over 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jill P. Buyon, Principal Investigator — Hospital for Joint Diseases
Locations (4):
- United States (4):
  - Yale University Medical Center, New Haven, Connecticut
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Hospital for Joint Diseases, New York, New York
  - New York University Medical Center, New York, New York

REFERENCES:
- [Background] Saleeb S, Copel J, Friedman D, Buyon JP. Comparison of treatment with fluorinated glucocorticoids to the natural history of autoantibody-associated congenital heart block: retrospective review of the research registry for neonatal lupus. Arthritis Rheum. 1999 Nov;42(11):2335-45. doi: 10.1002/1529-0131(199911)42:113.0.CO;2-3. PMID 10555029
- [Background] Glickstein JS, Buyon J, Friedman D. Pulsed Doppler echocardiographic assessment of the fetal PR interval. Am J Cardiol. 2000 Jul 15;86(2):236-9. doi: 10.1016/s0002-9149(00)00867-5. No abstract available. PMID 10913494
- [Background] Buyon JP, Waltuck J, Kleinman C, Copel J. In utero identification and therapy of congenital heart block. Lupus. 1995 Apr;4(2):116-21. doi: 10.1177/096120339500400207. PMID 7795614
- [Background] Copel JA, Buyon JP, Kleinman CS. Successful in utero therapy of fetal heart block. Am J Obstet Gynecol. 1995 Nov;173(5):1384-90. doi: 10.1016/0002-9378(95)90621-5. PMID 7503173
- [Background] Askanase AD, Friedman DM, Copel J, Dische MR, Dubin A, Starc TJ, Katholi MC, Buyon JP. Spectrum and progression of conduction abnormalities in infants born to mothers with anti-SSA/Ro-SSB/La antibodies. Lupus. 2002;11(3):145-51. doi: 10.1191/0961203302lu173oa. PMID 11999879
- [Background] Friedman DM, Rupel A, Glickstein J, Buyon JP. Congenital heart block in neonatal lupus: the pediatric cardiologist's perspective. Indian J Pediatr. 2002 Jun;69(6):517-22. doi: 10.1007/BF02722656. PMID 12139139
- [Background] Friedman D, Buyon J, Kim M, Glickstein JS. Fetal cardiac function assessed by Doppler myocardial performance index (Tei Index). Ultrasound Obstet Gynecol. 2003 Jan;21(1):33-6. doi: 10.1002/uog.11. PMID 12528158
- [Background] Askanase A, Friedman D, Glickstein J, Kim M, Buyon J. Potential Therapeutic window from normal heart rate (NHR) to advanced heart blcok and early detection of firts degree block by echocardiographic measurement of the mechanical PR interval. Arthritis Rheum. 2002; 46(suppl);5321.
- [Background] Buyon JP, Clancy RM. Neonatal lupus: review of proposed pathogenesis and clinical data from the US-based Research Registry for Neonatal Lupus. Autoimmunity. 2003 Feb;36(1):41-50. doi: 10.1080/0891693031000067340. PMID 12765470
- [Background] Buyon JP, Clancy RM. Neonatal lupus syndromes. Curr Opin Rheumatol. 2003 Sep;15(5):535-41. doi: 10.1097/00002281-200309000-00003. PMID 12960477
- [Background] Buyon JP, Hiebert R, Copel J, Craft J, Friedman D, Katholi M, Lee LA, Provost TT, Reichlin M, Rider L, Rupel A, Saleeb S, Weston WL, Skovron ML. Autoimmune-associated congenital heart block: demographics, mortality, morbidity and recurrence rates obtained from a national neonatal lupus registry. J Am Coll Cardiol. 1998 Jun;31(7):1658-66. doi: 10.1016/s0735-1097(98)00161-2. PMID 9626848
- [Background] Friedman D, Duncanson Lj, Glickstein J, Buyon J. A review of congenital heart block. Images Paediatr Cardiol. 2003 Jul;5(3):36-48. PMID 22368629
- [Result] Friedman DM, Kim MY, Copel JA, Davis C, Phoon CK, Glickstein JS, Buyon JP; PRIDE Investigators. Utility of cardiac monitoring in fetuses at risk for congenital heart block: the PR Interval and Dexamethasone Evaluation (PRIDE) prospective study. Circulation. 2008 Jan 29;117(4):485-93. doi: 10.1161/CIRCULATIONAHA.107.707661. Epub 2008 Jan 14. PMID 18195175